CLINICAL TRIAL: NCT06884072
Title: A Phase 1, Open-label, Randomized, Single Dose, 2-Treatment, 2-Sequence, 2-Period Crossover Study to Evaluate the Effect of a High-fat Meal on the Exposures of Pimicotinib Capsule in Healthy Subjects
Brief Title: A Study to Evaluate the Effect of a High-fat Meal on the Exposure of Pimicotinib Capsule in Healthy Subjects
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Abbisko Therapeutics Co, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ABSK021-111
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A: Pimicotinib 50mg (2x25mg) - High - fat Meal First, Then Fasting (Experimental): Subjects in Sequence A will be administered a single oral dose of 50 mg Pimicotinib capsules (2 x 25 mg) in a post-high-fat meal state on Day 1 of Period 1, and a single oral dose of 50 mg Pimicotinib capsules (2 x 25 mg) in a fasting state on Day 1 of Period 2.
  Interventions: Drug: Pimicotinib capsule
- Sequence B: Pimicotinib 50mg (2x25mg) - Fasting First, Then High - fat Meal (Experimental): Subjects in Sequence B will receive a single oral dose of 50 mg pimicotinib capsules (2 x 25 mg) in a fasting state on Day 1 of Period 1, and a single oral dose of 50 mg pimicotinib capsules (2 x 25 mg) in a post-high-fat meal state on Day 1 of Period 2.
  Interventions: Drug: Pimicotinib capsule

INTERVENTIONS:
Drug: Pimicotinib capsule — Pimicotinib capsule

SUMMARY:
This is a study to evaluate the impact of a high - fat meal on the exposure of Pimicotinib capsules in healthy subjects. It is planned to recruit 16 healthy subjects and randomly and equally assign them to either Study Sequence A or Study Sequence B. Subjects in Sequence A will take a single 50 - milligram oral dose of Pimicotinib capsules in a post - high - fat - meal state during Phase 1. Subjects in Sequence B will take a single 50 - milligram oral dose of Pimicotinib capsules in a fasting state during Phase 1 and then receive cross - over administration in Phase 2. In total, blood samples will be collected at 34 time points for pharmacokinetic (PK) analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects aged 18 to 50 years (inclusive) at screening;
2. Weight ≥ 50.0 kg (male) or ≥ 45.0 kg (female);
3. Normal or abnormal but not clinically significant results in medical history, physical examination, clinical laboratory tests and other relevant examinations as assessed by the investigator at Screening;
4. Male or female subjects of childbearing potential must agree to use effective methods of contraception during the study and within 6 months after the last dose of investigational product;
5. Willing to participate in this study, understand the study procedures and sign the informed consent form prior to screening; willing to comply with the study procedures.

Exclusion Criteria:

1. Past or current medical history of chronic or severe conditions in cardiovascular, respiratory, blood, liver, kidney, gastrointestinal, endocrine or nervous systems;
2. Known or persistent mental disorders;
3. Past history of gastric or intestinal surgery, or other operations;
4. Dysphagia and inability to take the investigational product orally;
5. Intolerant to venipuncture, difficult to collect blood samples, and fear of needle sickness and blood;
6. Known allergy to two or more kinds of foods and drugs; or allergic to pimicotinib or its excipients;and intolerance to dairy products;
7. History of infection within 30 days prior to screening;
8. Symptoms of fatigue and pyrexia within 2 weeks prior to screening;
9. Abnormal laboratory tests;
10. Positive result for either of the following tests: serum Hepatitis B Surface Antigen (HBsAg), Hepatitis C Virus (HCV) antibody, Human Immunodeficiency Virus (HIV) antibody, and treponema pallidum antibody;
11. Participated in any clinical studies of drugs as a study subject and received the study drug within 3 months prior to screening;
12. Previously participated in any other study related to pimicotinib and received pimicotinib;
13. Used strong inhibitors or inducers of CYP3A4 within 14 days prior to screening and at Screening or intending to use during the study;
14. Have special diet requirements and cannot accept to take a unified dietary;
15. Consumption of more than 14 units of alcohol per week within 3 months prior to signing the informed consent form, or a positive result for alcohol breath test on the day pre-dose, or unable to abstain from alcohol during the study;
16. Consumption of more than 5 cigarettes per day within 3 months prior to signing the informed consent form, or unable to abstain from tobacco products during the study;
17. Previous chronic consumption of excessive amount of tea, coffee, or caffeinated beverages or unable to abstain from caffeinated beverages during the study;
18. Known history of drug abuse or positive for drug abuse screening test;
19. Used over the counter or prescription drugs within 14 days prior to screening, or plan to use such drugs during the study;
20. Donated or lost > 400 mL of blood within 3 months prior to screening; received blood transfusions or used blood products within 2 months prior to screening;
21. Received vaccine within 2 months prior to screening, or plan to get vaccinated during the study;
22. Significant abnormalities and judged by the investigator as clinical significance in vital signs;
23. Heart rate-corrected QT interval prolongation;
24. Subjects involved in the design or conduct of this study and their immediate family members;
25. Subjects who, in the opinion of the investigator, are not suitable for enrollment or may not be able to complete the study for other reasons.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Cmax | Period 1& Period 2: pre-dose, postdose 15 minutes, 0.5 hour, 1 hour, 2 hours, 3 hours, 4 hours,5 hours, 6 hours, 8 hours, 24 hours, 48 hours, 96 hours, 120 hours, 144 hours, 192 hours and 240 hours.
  Peak concentration, the maximum observed plasma concentration of pimicotinib
AUC0-∞ | Period 1& Period 2: pre-dose, postdose 15 minutes, 0.5 hour, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 24 hours, 48 hours, 96 hours, 120 hours, 144 hours, 192 hours and 240 hours.
  Area under the plasma concentration-time curve of pimicotinib from time 0 to infinity, calculated as: AUC0-∞=AUClast +Clast/λz; Clast refers to the last measurable (non-BQL) plasma concentration of pimicotinib.
AUC last | Period 1& Period 2: pre-dose, postdose 15 minutes, 0.5 hour, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 24 hours, 48 hours, 96 hours, 120 hours, 144 hours, 192 hours and 240 hours.
  Area under the plasma concentration-time curve of pimicotinib from time 0 to the time of last measurable (non-BQL) concentration (calculated using the Linear Up Log Down trapezoidal method)

SECONDARY OUTCOMES:
t1/2 | Period 1& Period 2: pre-dose, postdose 15 minutes, 0.5 hour, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 24 hours, 48 hours, 96 hours, 120 hours, 144 hours, 192 hours and 240 hours.
  Elimination half-life
CL/F | Period 1& Period 2: pre-dose, postdose 15 minutes, 0.5 hour, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 24 hours, 48 hours, 96 hours, 120 hours, 144 hours, 192 hours and 240 hours.
  Total apparent clearance after a single oral dose
Vz/F | Period 1& Period 2: pre-dose, postdose 15 minutes, 0.5 hour, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 24 hours, 48 hours, 96 hours, 120 hours, 144 hours, 192 hours and 240 hours.
  Apparent volume of distribution after a single oral dose
AE | through study completion, an average of 26 days
  To evaluate the safety of a single oral administration of pimicotinib capsules in healthy subjects. The evaluation contents include adverse events (AE), serious adverse events (SAE), vital signs, physical examinations, electrocardiograms (ECG), and laboratory tests.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojiao Li, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China